CLINICAL TRIAL: NCT03037567
Title: Evaluation of a Commercial Program on Weight Loss and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-3421
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Weight Watchers plan (Experimental): Modified Weight Watchers Plan which includes a food plan, activity plan, group support and cognitive behavior modification. Weekly study-specific group meetings; electronic tools through iPhone app for 24 weeks.
  Interventions: Behavioral: Modified Weight Watchers plan

INTERVENTIONS:
Behavioral: Modified Weight Watchers plan — Weight Watchers is a structured lifestyle modification program that includes a food plan based on balanced diet and healthy eating, activity plan designed to promote progressive physical activity increase, group support and cognitive behavior modification. Participants attend weekly in-person group meetings led by a trained Weight Watchers meeting leader and have a suite of electronic tools available through an iPhone app.

SUMMARY:
The purpose of this study is to examine the acceptability and efficacy of a modified Weight Watchers program over 24 weeks. Assessments will be conducted at 0, 3, and 6 months.

DETAILED DESCRIPTION:
The following assessment measures will be taken at 0, 3, and 6 months:

Weight measurements. Weight will be taken according to the National Health and Nutrition Examination survey anthropometry procedures manual. Weight will be measured in kilograms to the nearest 0.1 kg using a calibrated digital scale (Tanita, Inc.) with participants in light clothing and no shoes. Two measurements will be taken. and if the measures differ by more than 0.2 kg, a third measure will be taken. An average of the closest two measures will be calculated and used for data entry.

Waist circumference. Waist circumference will be assessed at baseline, 3 and 6 months. Waist circumference will be taken according to the National Health and Nutrition Examination survey anthropometry procedures manual. Measurements will be taken to the nearest 0.1cm, at the top of the pelvis ilium (just above the hip bone) with a non-stretchable tape measure, without compressing the skin, at the end of normal expiration. Two measurements will be taken with a third if the first two do not fall within 0.5 cm.

Aerobic stamina. Aerobic stamina will be assessed using the 6 minute walk test. Distance traveled in meters (m) is the outcome.

Flexibility. Flexibility will be assessed with the Classic Sit and Reach Test and reported in inches less than or greater than reached on a 20 inch reference mark as measured on a yard stick placed between the legs.

Food Cravings. The Food Craving Inventory-II (FCI-II) is a validated self-report measure for general cravings and cravings for specific types of foods and will be completed at baseline, Months 3 and 6. Respondents rate the frequency of cravings since the last time they completed the survey for each of 33 food items using a five-point Likert scale (1, never; 2, rarely; 3, sometimes; 4, often; 5, always/almost every day). The FCI-II consists of 5 scales (sweets, high fats, carbohydrates/starches, fast food fats, and fruits & vegetables) that constitute the higher order construct of food cravings (the total score).

Happiness. The Oxford Happiness Questionnaire will be used to assess happiness at 0, 3, and 6 months. The OHQ is a validated self-report measure for broad personal happiness. Respondents rate 29 sentences on a 6 point Likert scale (1, strongly disagree; 6, strong agree).

Sleep. Participants will be asked to complete the Pittsburgh Sleep Quality Index (PSQI) to assess sleep quality and duration at 0, 3, 6. The PSQI is a validated self-report measure of sleep duration and sleep quality. The PSQI examines seven components of sleep quality retrospectively over a period of four weeks: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. The patient self-rates each of these seven areas of sleep. Scoring of answers is based on a 0-3 scale, whereby '3' reflects the negative extreme on the Likert scale. The global score is generated by summing up all seven component scores and ranges from 0 to 21, with higher values corresponding to reduced sleep quality.

Weight related quality of life. The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life. Respondents rate the degree to which their weight affects them on 31 items using a five-point Likert scale (1, never true; 2, rarely true; 3, sometimes true; 4, usually true; 5, always true). The IWQOL-Lite consists of 5 scales (physical function, self-esteem, sexual life, public distress, and work).

Perceived Hunger. The Visual Analogue Scale (VAS) measures sensations that range across a continuum of values and cannot be easily directly measured. Operationally, the VAS is a horizontal line measuring exactly 100 mm in length, anchored by word descriptors (i.e., Not at all hungry, Extremely hungry) at each end. Participants will be asked to complete a three item VAS by placing a mark on the line at the point they feel represents their response to the question.

Program Satisfaction. The Satisfaction Survey is a self-administered survey with 25 items scored on a 5-point Likert scale. This measure will be completed at only at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 43 kg/m²
* Ability to read and speak English
* All ethnic groups will be recruited
* Self-report desire to lose weight and willing to follow study recommendations
* Use of an iPhone with iOS 8.0 or later for use on a daily basis, and basic app skills
* Have access to the internet via a computer, and basic computer skills

Exclusion Criteria:

* Currently following a commercial weight-loss program (including Weight Watchers) or who followed a weight loss program in the previous 6 months or who were members of Weight Watchers within the past 12 months
* Another member of the household participating in the study.
* Pregnant or nursing, or planning on becoming pregnant over the next 9 months.
* Planning to relocate in the next 9 months
* Involvement in another research study that would interfere with participation in this study
* Excessive alcohol intake or dependence
* Recent weight loss of ≥ 5 kg in the previous 6 months.
* Report health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., orthopedic limitations, heart problems, history or heart attack or stroke)
* History of clinically diagnosed eating disorder.
* Untreated thyroid disease or and changes in dose or type of thyroid medication over previous 6 months
* Chronic/inflammatory gastrointestinal disorders (Irritable Bowel Syndrome acceptable)
* Taking any prescription medication with known effects on appetite or weight
* Previous surgical procedure for weight loss.
* Major surgery within the previous 6 months.
* Resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >100 mmHg
* Diuretic use over 1.5mg per day
* Diagnosis of type 1 or type 2 diabetes
* Presence of implanted cardiac defibrillator or pacemaker.
* History of presence of cancer within past 5 years or current treatment for cancer (completely resected basal or squamous cell carcinoma acceptable if treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Weight Change | 0 - 6 months
  Mean Change in body weight (kg) Body weight will be assessed on a calibrated digital scale and recorded to the nearest 0.1 kg.

SECONDARY OUTCOMES:
Achieving a weight loss of 5% or more | 0 - 6 months
  % participants achieving a weight loss of 5% initial body weight or more
Achieving a weight loss of 5% or more | 0 - 3 months
  % participants achieving a weight loss of 5% initial body weight or more
Weight Change | 0 - 3 months
  Mean Change in body weight (kg)
Waist circumference change (cm) (mean) | 0 - 3 months
  Waist circumference will be measured at the iliac crest
Waist circumference change (cm) (mean) | 0 - 6 months
  Waist circumference will be measured at the iliac crest
Relationship between fitness, flexibility and psychosocial measures with weight change | 0 - 6 months
  The relationship between weight change and any of these measures will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No